CLINICAL TRIAL: NCT05176964
Title: Combined Chemotherapy and Tislelizumab With Preoperative Split-course Hypofraction Radiotherapy for Locally Advanced Rectal Cancer:Study Protocol of a Prospective, Single-arm Phase II Trial
Brief Title: Chemotherapy and Tislelizumab With Split-course HFRT for Locally Advanced Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Benhua Xu, Director, Fujian Medical University Union Hospital
Other Study IDs: FujianUnionH-HFRT
Record Dates: First submitted 2021-11-30; First posted 2022-01-04 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Rectal Cancer; Radiation Oncology
Keywords: chemotherapy; tislelizumab; split-course hypofraction radiotherapy; locally advanced rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; tislelizumab; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, tumor tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HFRT with concurrent chemotherapy and immunotherapy: CAPOX chemotherapy plus tislelizumab treatment plus split-course HFRT
  Interventions: Radiation: split-course HFRT; Drug: CAPOX chemotherapy; Drug: Tislelizumab

INTERVENTIONS:
Radiation: split-course HFRT — 7Gy/F, d7, q3w, 5 cycles
  Other Names: hypofraction radiotherapy
Drug: CAPOX chemotherapy — CAPOX chemotherapy will commence on day 1 for each of six cycles: oxaliplatin 130 mg/m^2 intravenous infusion on day 1,followed by capecitabine 1000 mg/m^2 administered orally twice daily on day 1 to 14 of a 21-day cycle.
  Other Names: oxaliplatin and capecitabine
Drug: Tislelizumab — Tislelizumab 200 mg intravenous infusion on day 1 of each 21-day cycle for each of six cycles.
  Other Names: immunotherapy

SUMMARY:
The question of how to administer adequate chemotherapy and immunotherapy to synchronise hypofraction radiotherapy （HFRT） treatment strategy to maximise the benefits of neoadjuvant therapy for the improved prognosis of patients with locally advanced rectal cancer (LARC).We aimed to study whether chemotherapy and tislelizumab plus split-course HFRT results in better outcomes in LARC patients.

DETAILED DESCRIPTION:
Prior to analyzing continuous variables, the statistical normality of the data will be determined. The differences between the main variables will be compared by using the analysis of variance. A comparison of data on categorical variables will be carried out by χ2 tests or Fisher's exact tests. The OS and PFS was estimated using the Kaplan-Meier method. PFS and OS will be compared using the log-rank test. In cases where variables must be adjusted, we will use the proportional hazard Cox regression model. P values for all analyses will be based on using a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve patients with operable locally advanced cancer (LARC, T3-4 and/or N+)
* Pathologically diagnosed as rectal adenocarcinoma
* Male or non-pregnant female
* Age: 18-70 years old
* Hematology examination：I. White blood cell count ≥4×10^9/L;II. Neutrophils ≥1.5×10^9/L;III. Platelet count ≥100×10^9/L;IV. Hemoglobin ≥9g/L
* Blood biochemical examination: total bilirubin, AST, ALT≤2.0×upper limit of normal; creatinine≤1.5×upper limit of normal
* Functional status: ECOG score 0-1 points or KPS score ≥70 points
* Obtain the patient's informed consent

Exclusion Criteria:

* Pathologically diagnosed as non-adenocarcinoma
* Age> 70 years old
* Patients with recurrence and distant metastasis
* Have a history of other malignancies
* Have had radiotherapy and/or chemotherapy
* Pregnant or breastfeeding women
* Mentally disordered
* Patients with severe heart, liver, and kidney damage
* Non-compliance or the investigator believes that the patient cannot complete the entire trial treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hosptal in-patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response(pCR) | 1 year
  pCR is defined as no residual tumor in the surgical specimen.

SECONDARY OUTCOMES:
3-year disease-free survival | 2 years
  the time from randomization to disease recurrence or patient death due to disease progression.
local recurrence rate | 3 years
  It's defined as disease-free proximal, distal and circumferential margins.And its progression was defined as an increase in tumor size.
overall survival(OS) | 5 years
  It's defined as the time after the first dose of study therapy to death from any cause.
Sphincter-sparing surgery rate | 1 year
  sphincter-sparing surgery rate
R0 Resection Rate(R0-R) | 1 year
  It's defined as the percentage of patients undergoing resection, defined as a tumour-free resection margin.
predictive biomarkers andquality of life(QoL) | 3 years
  Objective condition index include subjective perception index objective condition index and subjective perception index.

CONTACTS AND LOCATIONS:
Overall Officials: Benhua Xu, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Zheng R, Wang BS, Li Z, Chi P, Xu B. Combining chemotherapy and tislelizumab with preoperative split-course hypofraction radiotherapy for locally advanced rectal cancer: study protocol of a prospective, single-arm, phase II trial. BMJ Open. 2023 Mar 16;13(3):e066976. doi: 10.1136/bmjopen-2022-066976. PMID 36927585